CLINICAL TRIAL: NCT00768352
Title: An Educational Intervention for Optimizing Adolescent Mental Health Screening Skills and Treatment in Pediatric Residency
Brief Title: Educational Intervention for Optimizing Adolescent Mental Health Screening and Treatment in Pediatric Residency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Capt Shana Hansen, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: C.2008.017e
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Mental Health
Keywords: Pediatric; Resident; Depression; Screening; Substance Abuse; Pediatric Resident knowledge of mental health topics; Pediatric Resident current practices for screening and treating mental health disorders; Pediatric Resident mental health care competency
MeSH Terms: conditions — Psychological Well-Being; Depression; Substance-Related Disorders | interventions — Early Intervention, Educational

ARMS (1):
- Education Intervention (Other)
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — An educational intervention which will consist of a standardized PowerPoint presentation that will cover general mental health topics such as depression and substance abuse. The presentation will also include discussion of common and validated mental health screening and assessment tools, as well as how to use these tools in a clinical setting. An educational packet will be provided to the residents and will include the screening tools, information on motivational interviewing and the behavioral stages of change, information on common medications prescribed for mental health disorders, and a bibliography of reputable resources for mental health topics.

SUMMARY:
The purpose of this study is: 1) to assess pediatric resident knowledge of adolescent mental health; 2) to assess pediatric resident comfort level for screening, assessing, and treating mental health disorders in adolescents, and; 3) to evaluate pediatric resident current practices for adolescent mental health screening, assessment, and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Residents
* Adolescent Rotation

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Do pediatric residents lack an adequate knowledge base for screening, assessing, and treating mental health disorders in adolescents? | Feb 2008-June 2009

SECONDARY OUTCOMES:
Are pediatric residents are comfortable with screening, assessing, and treating adolescent mental health disorders. Do pediatric residents use validated verbal or written mental health screening and assessment tools. | Feb 2008-June 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army medical Center, Fort Sam Houston, Texas, United States